CLINICAL TRIAL: NCT05258968
Title: Effectiveness of the Injeti Self-Esteem Model (ISEM) for Improving Self-esteem Among University
Brief Title: Injeti Self-Esteem Model and University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5210395
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Self Esteem
Keywords: Self Esteem; Relationships; University students

STUDY DESIGN:
Intervention Model Description: University students will be recruited to participate in 1 educational session on the Injeti Self Esteem Model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Session on the Injeti Self Esteem Model (Experimental): The participant will participate in a 1 hour educational session on the Injeti Self Esteem model.
  Interventions: Other: Education on the Injeti Model of Self-Esteem

INTERVENTIONS:
Other: Education on the Injeti Model of Self-Esteem — 1 hour educational session

SUMMARY:
The purpose of this study is to explore the effectiveness of the Injeti Self-Esteem Model (ISEM) with a psychoeducational therapy intervention for improving self-esteem among university students. To explore the effectiveness of the ISEM (see Appendix A), investigators are utilizing a mixed method study design to acquire both quantitative and qualitative data to view effectiveness through measurable outcomes and personal experience. The intervention will involve a 1-hour session, which will include administration of the ISEM.

DETAILED DESCRIPTION:
To explore the effectiveness of the ISEM investigators are utilizing a mixed-method study design to acquire both quantitative and qualitative data to view effectiveness through measurable outcomes and personal experience. Quantitative data will be gathered through standardized assessments, questionnaires, and demographic information. Qualitative information will be gathered through two interviews.

Pre-intervention data collection will include a Demographic Questionnaire, Rosenberg Self-Esteem Scale (RSES), and the Adverse Childhood Experience Questionnaire (ACE). The intervention itself will involve a 50-minute session consisting of the administration of the ISEM. All researchers will be trained to administer the ISEM by the Principal Investigator. After the intervention, data collection will involve two semi-structured interviews (SSI 1 and 2) that each require a completion of the RSES.

Inclusion/Exclusion Criteria.

Participants will include up to 150 students from varying universities throughout the Inland Empire ranging from 18-35 years of age. Participants must currently be enrolled as full-time or part-time students in an undergraduate or graduate program. English fluency in all areas (reading, writing, speaking, comprehension) will be required from all participants.

Investigators will recruit from each of the eight schools at Loma Linda University who have provided a signed Letter of Agreement (see Appendix B) using digital flyers via email communication. We will also recruit via snowballing.

The instruments we will use to collect data will include a Demographic Questionnaire, the Rosenberg Self-Esteem scale, the Adverse Childhood Experiences Questionnaire for Adults, and semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 35
* Must currently be enrolled as full-time or part-time students in an undergraduate or graduate program.
* English fluency in all areas (reading, writing, speaking, comprehension)

Exclusion Criteria:

* <18 or >35 years of age
* Does not meet student status
* Not fluent in English

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Self-Esteem | Change between baseline and 2 weeks post educational session
  The Rosenberg Self Esteem Scale is a10-item self-reported questionnaire designed to measure self-esteem. It includes 10 statements related to a person's feelings of self-worth or self-acceptance. A four-point scale ranging from "strongly agree" to "strongly disagree" is used to answer the questions (Rosenberg Self-Esteem Scale, n.d). The RSES is a reliable instrument as indicated by its Guttman scale coefficient of reproducibility of 0.92, which indicates excellent internal consistency. Test-retest reliability has correlations of 0.85 and 0.88 over a 2-week period, which indicates appropriate stability. The validity of the RSES is demonstrated by its concurrent, predictive, and constructive validity using known groups. The RSES correlates significantly with other measures of self-esteem such as the Coopersmith Self-Esteem Inventory as well as with the predicted direction of measures of depression and anxiety (Rosenberg, 2006).
Level of knowledge assessment | Change between 1 week Post educational session and 1 month post educational session.
  This semi-structured 15 minute interview will be completed after the educational session on the ISEM at two different time periods to gain an understanding of the participants perspective of how the knowledge has or has not been beneficial.

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Injeti, OTD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Information shared would relate to de-identified data analyzed for publication with our fellow researchers.
Supporting Information: SAP
Time Frame: After data collection.